CLINICAL TRIAL: NCT01096212
Title: A Multi-center, Open-Label, Randomized, Active-controlled, Parallel, Phase 4 Clinical Trial to Assess the Efficacy and Safety of Sevofran in Patients Scheduled for Elective Surgery Under General Anesthesia
Brief Title: Efficacy and Safety of Sevofran in Patients Scheduled for Elective Surgery Under General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: National Clinical Research Coordination Center, Seoul, Korea (Other Government)
Responsible Party: Gyu-Jeong Noh / Professor & Chairperson, Department of Clinical Pharmacology and Therapeutics, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asan Medical Center_sevofran_1
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: General Anesthesia; Sevoflurane; Generic Drugs
Keywords: Efficacy; Minimum alveolar concentration; Safety; Sevoflurane
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- generic sevoflurane (Experimental)
  Interventions: Drug: generic sevoflurane
- origianl sevoflurane (Active Comparator)
  Interventions: Drug: original sevoflurane

INTERVENTIONS:
Drug: original sevoflurane — Sevoflurane content: 99.9985%, compound A: 4.6 ppm, water content (sample was opened, sealed and stored for 2 weeks): 0.072% w/v
  Other Names: Sevorane® (Abott Korea Ltd, Seoul, Korea)
  Arms: origianl sevoflurane
Drug: generic sevoflurane — Sevoflurane content: 99.99%, compound A: 3.8 ppm, water content (sample was opened, sealed and stored for 2 weeks) : 0.044% w/v
  Other Names: Sevofran® (Hana Pharmacy, Co. Ltd, Seoul, Korea)
  Arms: generic sevoflurane

SUMMARY:
Sevoflurane is currently being used in more than 100 countries worldwide with an estimated 100 million operations having been performed using sevoflurane as a general anesthetic. After the expiry of the patent on sevoflurane as a pharmaceutical drug, a generic product (Sevofran®; Hana pharmacy, Co. Ltd, Seoul, Korea) has been launched. The aims of this study were to investigate the efficacy (mean minimum alveolar concentration), recovery characteristics (time to recovery of consciousness (ROC) and recovery, and BIS values at ROC and orientation), and safety (incidence and severity of adverse events) of generic sevoflurane in patients undergoing elective surgery.

DETAILED DESCRIPTION:
Patients were randomly allocated to experimental group (generic sevoflurane) and active comparator group (original sevoflurane). Once in the operating room, patients were monitored with electrocardiography, non invasive blood pressure, pulse oximetry (Datex-Ohmeda S/5, Planar Systems, Inc., Beaverton, OR, USA) and BIS (Aspect 2000, Aspect Medical Systems, Inc., Newton, MA, USA).

Anesthesia was induced with fentanyl (2 μg/kg) and propofol (2mg/kg). When patients were unconscious, original or generic sevoflurane was administered. Tracheal intubation was facilitated by administering rocuronium 0.6 mg/kg. The lungs of the patients were then ventilated with oxygen in air (1:2), and the ventilation rate was adjusted to maintain the end-tidal carbon dioxide partial pressure between 35 and 45 mmHg. The concentrations of carbon dioxide, sevoflurane, and oxygen were measured continuously using an infrared anesthetic gas analyzer (Datex-Ohmeda S/5, Planar Systems, Inc., Beaverton, OR, USA), which was calibrated before anesthesia for each patient using a standard gas mixture.

The inspired concentration of sevoflurane was adjusted to maintain BIS values < 60 and stable haemodynamics (systolic arterial pressure (SAP) > 80 mmHg and heart rate (HR) > 45 beats/min). Also, it was titrated to prevent signs of inadequate anesthesia (sweating, facial flushing, movement and swallowing, HR > 90 beats/min without evidence of hypovolemia, and a 15 mmHg increase in SAP, compared with baseline SAP). Fentanyl 1 μg/kg was given if needed to resolve of signs of inadequate anesthesia.

Concentration of compound A, formaldehyde, and methadone were measured at preset interval: 30, 60, 90, 120, 150, 180 min after administration of sevoflurane. Blood and urine samples were taken at preset interval for analyzing concentration of inorganic fluoride: 1 hr after administration of sevoflurane and every 2 hr during maintenance of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery under general anesthesia
* American Society Anesthesiologists Physical Status (ASA PS) 1 or 2
* Aged 19 years or above

Exclusion Criteria:

* ASA PS 3 or above
* aged under 19 years
* Contraindications against the use of sevoflurane
* Abnormal laboratory finding with clinical significance
* Evidence of pregnancy
* History of alcohol or drug abuse
* Hemoglobin < 11 mg/dl
* Neurological or psychiatric disease
* Unable or unwilling to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Comparison of mean minimum alveolar concentration between original and generic sevoflurane | During mainenance of anesthesia under general anesthesia
  Minimum alveolar concentration was determined by end-tidal sevoflurane concentrations. Mean MAC was calculated as following equation,
  Mean MAC = (MAC * hour) / (maintenance time from administration of hypnotic agent (propofol) for acquring loss of consciousness to extubation)

SECONDARY OUTCOMES:
Comparison of secondary efficacy and safety endpoints between two inhalation agents | During maintenance of anesthesia under general anesthesia
  Secondary efficacy and safety characteristics include following items.
  1. Anesthesia exposure: MAC * hour [Time frame: maintenanane period of anesthesia]
  2. Bispectral index, BIS [Time frame: time to recovery of consciousnessn, time to recovery of orientation]
  3. Adverse event [Time frame: maintenanane period of anesthesia]
  4. Incidence and severity of postopertive nausea and vomiting [Time frame: 24 hours postoperatively]
  5. Concentrations of compound A, formaldehyde, methanol [Time frame: 30, 60, 90, 120, 150, 180 min after sevoflurane administration]

CONTACTS AND LOCATIONS:
Overall Officials: Gyu Jeong Noh, M.D. & Ph.D., Study Chair — Department of Clinical Pharmacology and Therapeutics, Asan Medical Center, University of Ulsan College of Medicine; Sang Seok Lee, M.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, Sanggye-Paik Hospital, College of Medicine, Inje University
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Sanggye-Paik Hospital, Seoul

REFERENCES:
- [Derived] Byon HJ, Choi BM, Bang JY, Lee EK, Lee SS, Noh GJ. An Open-label Comparison of a New Generic Sevoflurane Formulation With Original Sevoflurane in Patients Scheduled for Elective Surgery Under General Anesthesia. Clin Ther. 2015 Apr 1;37(4):887-901. doi: 10.1016/j.clinthera.2015.01.012. Epub 2015 Feb 16. PMID 25697421